CLINICAL TRIAL: NCT04507555
Title: Pharmacist Guided Pre-emptive Pharmacogenetic Testing in Antidepressant Therapy
Acronym: PrePGx
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: PD Dr. med. Thorsten Mikoteit (Other)
Collaborators: Psychiatrische Dienste Solothurn (Unknown); Privatklinik Wyss (Unknown); Luzerner Psychiatrie AG (Unknown); Psychiatrische Universitätsklinik Zürich (Unknown)
Responsible Party: Sponsor-Investigator, PD Dr. med. Thorsten Mikoteit, Deputy Head Physician Division Psychiatry, University of Basel
Organization: University of Basel (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PrePGx_ex20Mikoteit
Record Dates: First submitted 2020-08-04; First posted 2020-08-11 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention (Experimental)
  Interventions: Procedure: Pharmacist-guided pharmacogenetic (PGx) testing for antidepressant selection and dosing
- Standard Care (Active Comparator)
  Interventions: Procedure: Standard care antidepressant selection and dosing
- Observational (No Intervention)

INTERVENTIONS:
Procedure: Pharmacist-guided pharmacogenetic (PGx) testing for antidepressant selection and dosing — The study intervention is the service of pharmacist guided pre-emptive PGx testing to support clinical decision making for antidepressant selection and dosing.
  This service involves genotyping and thereof evidence-based genotype interpretation commercially offered as Stratipharm® (humatrix AG, Pfungstadt Germany, https://www.stratipharm.de). Furthermore, clinical pharmacists will process and evaluate the results from PGx testing (Stratipharm®) in context of the individual patient medication history as well as current co-medication and forward an individualized recommendation for antidepressant selection and dosing to the treating psychiatrist.
  Arms: Intervention
Procedure: Standard care antidepressant selection and dosing — Selection and dosing of the new antidepressant pharmacotherapy will be determined by the treating investigator alone, according to current standard of care considering clinical factors only.
  Arms: Standard Care

SUMMARY:
In this study at the Solothurn Psychiatric Clinic, the investigators compare the effectiveness and tolerability of antidepressant pharmacotherapy in three groups. In the intervention group, the physician selects and doses the medication for depression based on a pharmacogenetic examination conducted by a clinical pharmacist. In the standard group, the treating physician selects and doses the antidepressant drug without the support of genetic testing, in accordance with current standard practice. If after the first week of hopsitalization no adjustment to a new antidepressant is necessary, the investigators will monitor the progress of these patients until they leave the clinic in an observational arm. The drugs used are all approved in Switzerland for the treatment of depression. Classification into the intervention or standard group is made randomly after the first week of hospitalisation, if the treating physician deems it necessary to change or readjust the antidepressant pharmacotherapy. The probability of allocation to one of the two study groups is 50%. All study participants will be hospitalized for at least five weeks and monitored until they leave the clinic. In total, it is planned to include and examine 95 patients each into the intervention and standard group.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Diagnosis unipolar moderate or severe depressive episode or recurrent depressive disorder (ICD10: F32.1/32.2/33.1/33.2)
* HAM-D17 ≥ 17

Exclusion Criteria:

* Acute suicide risk
* Psychotic symptomatology
* Other acute serious psychiatric disorder other than depression
* Excessive consumption of alcohol and/or drugs
* Severe acute - or severe chronic somatic diseases
* Pregnant / lactating women
* Under current treatment with fluoxetine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
rate of response to the antidepressant therapy at the end of week 4 | 28 days
  response is determined as a reduction in the Hamilton Depression (HAM-D17) Scale score of at least 50 % of the baseline value

SECONDARY OUTCOMES:
Time to response | 28 days
  time span from start of antidepressant pharmacotherapy until first assessed response (= HAM-D17 reduction of at least 50 % compared to baseline
Remission rate | 28 days
  17 item Hamilton rating scale for Depression (HAM-D17) score ≤ 8
Overall change in 17 item Hamilton rating scale for Depression (HAM-D17) from baseline to week 4 | 28 days
  minimum value: 0, maximum value: 52 ; higher scores mean worse outcome
Time till discharge | assessed up to 3 month
  time span from admission (randomization) to discharge from inpatient treatment
Patient depression self-rating | 28 days
  two weekly assessment with Beck's Depression Inventory questionnaire (BDI-II)
Side effect measure (self-rated frequency, intensity and burden of side effects, FIBSER score) | 28 days
  weekly assessment, minimum value: 0, maximum value: 18 ; higher scores mean worse outcome
Number of adverse events related to antidepressant pharmacotherapy | 28 days
  severity grading ≥ 2 (using CTCAE version 5.0) and causality to antidepressant pharmacotherapy assessed as possible, probable or definite

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Mikoteit, PD Dr. med., Principal Investigator — Psychiatrische Dienste Solothurn
Locations (4):
- Switzerland (4):
  - Privatklinik Wyss, Münchenbuchsee, Canton of Bern
  - Psychiatrische Dienste Solothurn, Solothurn, Canton of Solothurn
  - Luzerner Psychiatrie AG, Sankt Urban
  - Psychiatrische Universitätsklinik Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stauble CK, Lampert ML, Allemann S, Hatzinger M, Hersberger KE, Meyer Zu Schwabedissen HE, Imboden C, Mikoteit T. Pharmacist-guided pre-emptive pharmacogenetic testing in antidepressant therapy (PrePGx): study protocol for an open-label, randomized controlled trial. Trials. 2021 Dec 14;22(1):919. doi: 10.1186/s13063-021-05724-5. PMID 34906208